CLINICAL TRIAL: NCT02440191
Title: Postoperative Radiotherapy With Intensity-modulated Radiation Therapy (IMRT) Using Simultaneous Integrated Boost Versus 3-dimensional Conformal Radiotherapy (3D-CRT) in Early Breast Cancer: a Prospective Randomized Trial
Brief Title: 3DCRT vs. IMRT in Early Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jong Hoon Lee (Other)
Responsible Party: Sponsor-Investigator, Jong Hoon Lee, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KROG 15-03
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Radiation Toxicity
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3DCRT (Active Comparator): conventional 3-dimensional conformal radiotherapy on the breast, 50.4 Gy/28 fx and tumor bed boost, 9 Gy/5 fx will be irradiated for 6.5 weeks.
  Interventions: Radiation: 3DCRT
- IMRT (Intensity modulated radiotherapy) (Experimental): Intensity-modulated radiotherapy (IMRT) with simultaneous integrated boost (SIB) on the whole breast, 50.4 Gy/28 fx and tumor bed, 57.4 Gy/28 fx will be irradiated for 5.5 weeks.
  Unlike 3DCRT, concomittant boost technique is used in the IMRT arm.
  Interventions: Radiation: 3DCRT

INTERVENTIONS:
Radiation: 3DCRT — conventional radiotherapy

SUMMARY:
It has been not clinically determined whether TomoDirect was dosimetrically better than 3D-CRT for Asian patients with early breast cancer. Therefore, the objective of this study was to compare dosimetric parameters of TomoDirect and 3D-CRT in early breast cancer patients of an Asian cohort.

DETAILED DESCRIPTION:
In breast cancer patients, helical TomoTherapy is not a suitable option since the gantry continuously rotates around the patient, and this technique can deliver low dose radiation to lungs that is associated with an occurrence of radiation pneumonitis. To avoid this inefficiency of beam usage, a TomoDirect option using static gantry positions combined with simultaneous couch translation and dynamic collimator modulation has been developed. In a pilot study, TomoDirect seemed particularly well suited for postoperative irradiation in breast cancer patients. TomoDirect achieved an optimal target volume coverage and coincident adequate normal tissue sparing in a dosimetric study. Clinical studies of TomoDirect in breast cancer patients are scarce and have been assessed only in small and retrospective series. Thus, we undertook a prospective study on the technical feasibility and toxicity of TomoDirect in breast cancer patients who received postoperative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed breast cancer after breast-conserving surgery
2. pT1-2N0
3. no evidence of distant metastasis
4. no previous malignancy
5. patient age, 20 - 80 years
6. Karnofsky performance score ≥ 70
7. adequate bone marrow, liver, and renal function (leucocytes > 4,000/mm3, hemoglobin > 10 g/dL, platelets > 100,000/mm3; serum bilirubin < 1.5 mg/dL, serum transaminase < 2.5 times the upper normal limit; serum creatinine < 1.5 mg/dL).
8. completion of scheduled chemotherapy

Exclusion Criteria:

1. carcinoma in situ of breast
2. distant metastasis
3. mastectomy
4. male
5. both breast cancer

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-year

SECONDARY OUTCOMES:
Toxicity | acute (time frame: with 3 months after radiation) and late (time frame: up to 3 years after radiation), Participants will be followed for an expected average of 3 years.
  Acute toxicity within 3 months after radiotherpy and late toxicity thereafter up to 3 years will be followed up by physicians. Adverse effects of radiotherapy were assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0). Incidence of toxicity grade ≥ 2 was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hoon Lee, MD, Principal Investigator — St. Vincent's Hospital, The Catholic University of Korea
Locations (1):
- St. Vincent Hospital, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Capelle L, Warkentin H, Mackenzie M, Joseph K, Gabos Z, Pervez N, Tankel K, Chafe S, Amanie J, Ghosh S, Parliament M, Abdulkarim B. Skin-sparing helical tomotherapy vs 3D-conformal radiotherapy for adjuvant breast radiotherapy: in vivo skin dosimetry study. Int J Radiat Oncol Biol Phys. 2012 Aug 1;83(5):e583-90. doi: 10.1016/j.ijrobp.2012.01.086. Epub 2012 May 12. PMID 22580119
- [Derived] Choi KH, Ahn SJ, Jeong JU, Yu M, Kim JH, Jeong BK, Lee JH, Kim SH, Lee JH. Postoperative radiotherapy with intensity-modulated radiation therapy versus 3-dimensional conformal radiotherapy in early breast cancer: A randomized clinical trial of KROG 15-03. Radiother Oncol. 2021 Jan;154:179-186. doi: 10.1016/j.radonc.2020.09.043. Epub 2020 Sep 24. PMID 32980384